CLINICAL TRIAL: NCT02065986
Title: Pre-exposure Option for Reducing HIV in the UK: an Open-label Randomisation to Immediate or Deferred Daily Truvada for HIV Negative Gay Men.(PROUD)
Brief Title: Pre-exposure Option for Reducing HIV in the UK.(PROUD)
Acronym: PROUD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MRC [ycm] (Other Government)
Responsible Party: Sponsor-Investigator, MRC [ycm], Medical Research Council, Medical Research Council
Organization: Medical Research Council (Other Government)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2012-002373-56
Record Dates: First submitted 2014-02-16; First posted 2014-02-19 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: HIV
Keywords: HIV; Prevention; Truvada
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Immediate offer of Truvada-PrEP (Experimental): Immediate offer of Truvada (once daily tablet containing 300mg tenofovir disoproxil (TDF) and 200mg of emtricitabine (FTC)
  Interventions: Drug: Truvada (once daily tablet containing 300mg tenofovir disoproxil (TDF) and 200mg of emtricitabine (FTC)
- Arm B: Deferred (12m) offer of Truvada-PrEP (Other): Access to Truvada from 12 months after enrolment
  Interventions: Drug: Truvada (once daily tablet containing 300mg tenofovir disoproxil (TDF) and 200mg of emtricitabine (FTC)

INTERVENTIONS:
Drug: Truvada (once daily tablet containing 300mg tenofovir disoproxil (TDF) and 200mg of emtricitabine (FTC)

SUMMARY:
This study is looking at a new way to reduce the risk of catching HIV - Truvada-PrEP.

To find out whether a daily tablet, Truvada, can safely reduce the risk of gay men catching HIV, we need to do a large trial in which half the men do not receive Truvada for one year. We do not know if gay men at risk of HIV are interested in taking Truvada, and if they are, whether they would be willing to wait a year before they can take it. The reason it may not be safe, is that taking Truvada-PrEP may lead to an increase in risk behaviour. This could mean there was more chance of catching HIV and other infections.

As well as finding out if a large trial would be possible, this study will looks at other factors including:

* Whether people using PrEP change the number of partners they have sex with
* Whether people using PrEP change how often they use condoms
* Whether PrEP leads to higher rates of other sexually transmitted infections (STIs).

This information on changes in sexual activity over time is one of the most important aspects of the study, because we have never collected this before in the UK. This means we don't know what happens to people's sexual activity without PrEP! In October 2014 an interim analysis of the PROUD study data showed that pre-exposure prophylaxis (PrEP) was highly protective against HIV for gay men and other men who have sex with men (MSM) at high risk of infection. The PROUD Trial Steering Committee announced that participants on the deferred arm of the study, who had not yet started PrEP, should be offered the opportunity to begin PrEP ahead of schedule. As a result, we changed the study design and offered all enrolled participants the opportunity to access PrEP. All study participants will be followed up until study closure in October 2016

DETAILED DESCRIPTION:
Intervention and control groups:

Arm A: Immediate offer of Truvada-PrEP Arm B: Deferred (12m) offer of Truvada-PrEP

Method of randomisation:

Randomisation will be performed centrally using a computer algorithm based on random permuted blocks stratified by site.

ELIGIBILITY:
Inclusion Criteria:

* Born to male gender, age 18 years or more
* Previously attended the enrolling clinic on at least one occasion
* Completed a screen for HIV and STIs
* HIV negative by a routinely used assay within 4 weeks prior to or on the day of randomisation
* Reported unprotected anal intercourse (UAI) on more than one occasion within the 90 days prior to randomisation
* Likely, in the opinion of the volunteer, to have UAI in the next 90 days
* Willing and able to comply with the visit schedule throughout the follow-up period
* Willing and able to provide written informed consent

Exclusion Criteria:

* An acute viral illness that could be due to HIV seroconversion
* Any contraindications to Truvada according to the current package insert
* Treatment for hepatitis B infection indicated or ongoing
* Unlikely, in the opinion of the clinician, to comply with the randomised allocation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Time to accrual of 500 participants and Retention at 12 and 24 months from randomisation | 2 years

SECONDARY OUTCOMES:
HIV infections acquired between trial entry and 12 months, and between 12 and 24 months | 24months

CONTACTS AND LOCATIONS:
Locations (1):
- MRC Clinical Trials Unit, London, United Kingdom

REFERENCES:
- [Derived] Miltz A, Lampe F, McCormack S, Dunn D, White E, Rodger A, Phillips A, Sherr L, Sullivan AK, Reeves I, Clarke A, Gafos M. Prevalence and correlates of depressive symptoms among gay, bisexual and other men who have sex with men in the PROUD randomised clinical trial of HIV pre-exposure prophylaxis. BMJ Open. 2019 Dec 10;9(12):e031085. doi: 10.1136/bmjopen-2019-031085. PMID 31826890
- [Derived] Miltz AR, Lampe FC, Bacchus LJ, McCormack S, Dunn D, White E, Rodger A, Phillips AN, Sherr L, Clarke A, McOwan A, Sullivan A, Gafos M. Intimate partner violence, depression, and sexual behaviour among gay, bisexual and other men who have sex with men in the PROUD trial. BMC Public Health. 2019 Apr 25;19(1):431. doi: 10.1186/s12889-019-6757-6. PMID 31023281
- [Derived] McCormack S, Dunn DT, Desai M, Dolling DI, Gafos M, Gilson R, Sullivan AK, Clarke A, Reeves I, Schembri G, Mackie N, Bowman C, Lacey CJ, Apea V, Brady M, Fox J, Taylor S, Antonucci S, Khoo SH, Rooney J, Nardone A, Fisher M, McOwan A, Phillips AN, Johnson AM, Gazzard B, Gill ON. Pre-exposure prophylaxis to prevent the acquisition of HIV-1 infection (PROUD): effectiveness results from the pilot phase of a pragmatic open-label randomised trial. Lancet. 2016 Jan 2;387(10013):53-60. doi: 10.1016/S0140-6736(15)00056-2. Epub 2015 Sep 9. PMID 26364263